CLINICAL TRIAL: NCT05350345
Title: Safety Incident Reporting System for Students During Their Clinical Internship (SAFEST)
Acronym: SAFEST
Status: Completed | Type: Observational
Sponsor: Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana (Other)
Responsible Party: Principal Investigator, José Joaquín Mira Solves, University Professor (2012) with a position as Clinical Psychologist (1984) in Primary Care, Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana
Other Study IDs: UGP-21-215
Record Dates: First submitted 2022-04-22; First posted 2022-04-28 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Patient Safety
Keywords: Patient Safety; Safety Incident; Student; Report System
MeSH Terms: interventions — Root Cause Analysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Root-cause analysis — The first part of this study involves a report with a root-cause analysis done by the students. The second part is a gamification in which they have to evaluate each other and give feedback.
  Other Names: Gamification

SUMMARY:
Patient safety is a priority in Europe. The World Health Organization's World Alliance for Patient Safety has included incident reporting systems as indispensable tools for patient safety. These systems are widespread in healthcare facilities throughout Europe. While in some countries trainees in healthcare disciplines are able to report incidents, in others they are unable to do so. In many cases, they do not have adequate information about the reporting systems, there is low motivation to report, or there is a fear that reporting may lead to problems in their studies.

Until now, there have been no interventions designed and validated to achieve the objective of promoting incident reporting among students of health disciplines. Nor there were tools for these students to participate in the analysis of the causes of these incidents and in the identification of barriers to prevent their recurrence.

Researchers currently have tools from the digital world (artificial intelligence and gamification) whose application in this area can be useful for improving patient safety.

In this context, the investigators have developed an incident notification system aimed at students and trainees in order to familiarize this group with the notification process and thus contribute to improving patient safety. Students will be encouraged to participate with the incentive of earning Miguel Hernández University nanocourse credits or direct prizes. Once the notification is made, their role will be to evaluate and give feedback to notifications made by other peers, so they will get points. After finishing, those students with the most points will be rewarded with the prizes mentioned above.

ELIGIBILITY:
Inclusion Criteria:

* Students with Clinical Practices.

Exclusion Criteria:

-

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All students during their clinical internship can participate in this study.
Sampling Method: Non-Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2022-04-09 (Actual); Primary Completion 2023-11-08 (Actual); Study Completion 2023-11-08 (Actual)

PRIMARY OUTCOMES:
Root-cause analysis | 5 months
  An analysis of the causes of the problem will be carried out to try to prevent its recurrence in the future.

CONTACTS AND LOCATIONS:
Locations (1):
- Grupo ATENEA, Sant Joan d'Alacant, Alicante, Spain

REFERENCES:
- [Background] Donal, L. (2020). Patient Safety Incident Reporting and Learning Systems: Technical report and guidance. In World Health Organization.
- [Background] Scott, C.M., Lubritz, R.R., Graham, G.F. (2016). Adverse Events. In: Abramovits, W., Graham, G., Har-Shai, Y., Strumia, R. (eds) Dermatological Cryosurgery and Cryotherapy. Springer, London. https://doi.org/10.1007/978-1-4471-6765-5_47
- [Derived] Gil-Hernandez E, Carrillo I, Guilabert M, Bohomol E, Serpa PC, Ribeiro Neves V, Maluenda Martinez M, Martin-Delgado J, Perez-Esteve C, Fernandez C, Mira JJ. Development and Implementation of a Safety Incident Report System for Health Care Discipline Students During Clinical Internships: Observational Study. JMIR Med Educ. 2024 Jul 18;10:e56879. doi: 10.2196/56879. PMID 39024005